CLINICAL TRIAL: NCT02120456
Title: Safety and Efficacy of Escalating Doses of LEO 43204 Applied Once Daily for Two Consecutive Days on Approximately 250 cm2 on Trunk and Extremities in Subjects With Actinic Keratosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LP0084-1015
Record Dates: First submitted 2014-04-18; First posted 2014-04-22 (Estimated); Results first posted 2019-01-04 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2018-11

CONDITIONS: Actinic Keratosis
MeSH Terms: conditions — Keratosis, Actinic | interventions — LEO 43204

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- LEO 43204 (Experimental): Open-label, dose-escalation, 2-day treatment
  Interventions: Drug: LEO 43204
- LEO 43204 Dose 0.1% (Experimental): LEO 43204 dose 0.1% once daily for two consecutive days
  Interventions: Drug: LEO 43204
- LEO 43204 Dose 0.075% (Experimental): LEO 43204 dose 0.075% once daily for two days
  Interventions: Drug: LEO 43204
- Placebo (Placebo Comparator): Placebo once daily for two days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LEO 43204
  Arms: LEO 43204; LEO 43204 Dose 0.075%; LEO 43204 Dose 0.1%
Drug: Placebo
  Arms: Placebo

SUMMARY:
Part 1: To identify Maximum Tolerated Dose (MTD) levels of LEO 43204 after once daily treatment for two consecutive days

Part 2: To evaluate the efficacy of LEO 43204 in two doses after once daily treatment for two consecutive days compared to vehicle

ELIGIBILITY:
Inclusion Criteria:

* Part 1: Subjects with 5 to 20 clinically typical, visible and discrete AKs on the arm
* Part 2: Subjects with 5 to 20 clinically typical, visible and discrete AKs on the extremities or trunk

Exclusion Criteria:

* Location of the treatment area

  * within 5 cm of an incompletely healed wound
  * within 5 cm of a suspected basal cell carcinoma (BCC) or squamous cell carcinoma (SCC)
* Prior treatment with ingenol mebutate gel on the treatment area
* Lesions in the treatment areas that have:

  * atypical clinical appearance (e.g., hypertrophic, hyperkeratotic or cutaneous horns) and/or
  * recalcitrant disease (e.g., did not respond to cryotherapy on two previous occasions)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2014-05; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary Goldenberg, MD, Principal Investigator — Mount Sinai School of Medicine, Dermatology Faculty
Locations (21):
- United States (13):
  - Omni Dermatology, Phoenix, Arizona
  - Torrance Clinical Research Institute Inc., Lomita, California
  - Dermatology Cosmetic Laser Medical Associates of La Jolla, Inc., San Diego, California
  - Dermatology Associates and Research, Coral Gables, Florida
  - Leavitt Medical Associates of Florida, Ormond Beach, Florida
  - Deaconess Clinic, Inc., Evansville, Indiana
  - Hudson Dermatology, LLC, Evansville, Indiana
  - Indiana Clinical Trials Center, Plainfield, Indiana
  - DermAssociates, PC, Rockville, Maryland
  - Great Lakes Research Group, Inc., Bay City, Michigan
  - The Dermatology Group, P.C., Verona, New Jersey
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Pflugerville Dermatology Clinical Research Center, Inc., Pflugerville, Texas
- Canada (8):
  - Kirk Barber Research, Calgary, Alberta
  - Enverus Medical, Surrey, British Columbia
  - Skin Care Centre, Vancouver, British Columbia
  - Winnipeg Clinic Dermatology Research, Winnipeg, Manitoba
  - UltraNova Skincare, Barrie, Ontario
  - Dermatrials Research Incorporated, Hamilton, Ontario
  - The Guenther Dermatology Research Centre, London, Ontario
  - SKiN Centre for Dermatology, Peterborough, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Clinical Trials at LEO Pharma — https://www.leopharmatrials.com/en

RESULTS

PARTICIPANT FLOW:
Groups:
- Part 1: LEO 43204 Gel 0.018%: Once daily treatment for two consecutive days with LEO 43204 gel 0.018% on sun exposed area of 250 cm2 on the arm between wrist and shoulder.
- Part 1: LEO 43204 Gel 0.025%: Once daily treatment for two consecutive days with LEO 43204 gel 0.025% on sun exposed area of 250 cm2 on the arm between wrist and shoulder.
- Part 1: LEO 43204 Gel 0.037%: Once daily treatment for two consecutive days with LEO 43204 gel 0.037% on sun exposed area of 250 cm2 on the arm between wrist and shoulder.
- Part 1: LEO 43204 Gel 0.05%: Once daily treatment for two consecutive days with LEO 43204 gel 0.05% on sun exposed area of 250 cm2 on the arm between wrist and shoulder.
- Part 1: LEO 43204 Gel 0.075%: Once daily treatment for two consecutive days with LEO 43204 gel 0.075% on sun exposed area of 250 cm2 on the arm between wrist and shoulder.
- Part 1: LEO 43204 Gel 0.1%: Once daily treatment for two consecutive days with LEO 43204 gel 0.1% on sun exposed area of 250 cm2 on the arm between wrist and shoulder.
- Part 2: LEO 43204 Vehicle Gel: Once daily treatment for two consecutive days with LEO 43204 vehicle gel on sun exposed area of 250 cm2 on the extremities or trunk (except chest).
- Part 2: LEO 43204 Gel 0.075%: Once daily treatment for two consecutive days with LEO 43204 gel 0.075% on sun exposed area of 250 cm2 on the extremities or trunk (except chest).
- Part 2: LEO 43204 Gel 0.1%: Once daily treatment for two consecutive days with LEO 43204 gel 0.1% on sun exposed area of 250 cm2 on the extremities or trunk (except chest).
Period: Part 1 Open-label, Dose-escalation Phase
Arm/Group | Part 1: LEO 43204 Gel 0.018% | Part 1: LEO 43204 Gel 0.025% | Part 1: LEO 43204 Gel 0.037% | Part 1: LEO 43204 Gel 0.05% | Part 1: LEO 43204 Gel 0.075% | Part 1: LEO 43204 Gel 0.1% | Part 2: LEO 43204 Vehicle Gel | Part 2: LEO 43204 Gel 0.075% | Part 2: LEO 43204 Gel 0.1%
Started | 12 | 12 | 12 | 12 | 12 | 9 | 0 | 0 | 0
Completed | 12 | 12 | 12 | 12 | 12 | 9 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2 Double-blind Phase
Arm/Group | Part 1: LEO 43204 Gel 0.018% | Part 1: LEO 43204 Gel 0.025% | Part 1: LEO 43204 Gel 0.037% | Part 1: LEO 43204 Gel 0.05% | Part 1: LEO 43204 Gel 0.075% | Part 1: LEO 43204 Gel 0.1% | Part 2: LEO 43204 Vehicle Gel | Part 2: LEO 43204 Gel 0.075% | Part 2: LEO 43204 Gel 0.1%
Started | 0 | 0 | 0 | 0 | 0 | 0 | 32 | 60 | 63
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 30 | 60 | 62
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal of consent | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Unable to attend visit due to work | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Part 1: LEO 43204 Gel 0.018%: Once daily treatment for two consecutive days with LEO 43204 gel 0.018%
- Part 1: LEO 43204 Gel 0.025%: Once daily treatment for two consecutive days with LEO 43204 gel 0.025%
- Part 1: LEO 43204 Gel 0.037%: Once daily treatment for two consecutive days with LEO 43204 gel 0.037%
- Part 1: LEO 43204 Gel 0.05%: Once daily treatment for two consecutive days with LEO 43204 gel 0.05%
- Part 1: LEO 43204 Gel 0.075%: Once daily treatment for two consecutive days with LEO 43204 gel 0.075%
- Part 1: LEO 43204 Gel 0.1%: Once daily treatment for two consecutive days with LEO 43204 gel 0.1%
- Part 2: LEO 43204 Vehicle Gel: Once daily treatment for two consecutive days LEO 43204 vehicle gel
- Part 2: LEO 43204 Gel 0.075%: Once daily treatment for two consecutive days LEO 43204 gel 0.075%
- Part 2: LEO 43204 Gel 0.1%: Once daily treatment for two consecutive days LEO 43204 gel 0.1%
- Total: Total of all reporting groups
Arm/Group | Part 1: LEO 43204 Gel 0.018% | Part 1: LEO 43204 Gel 0.025% | Part 1: LEO 43204 Gel 0.037% | Part 1: LEO 43204 Gel 0.05% | Part 1: LEO 43204 Gel 0.075% | Part 1: LEO 43204 Gel 0.1% | Part 2: LEO 43204 Vehicle Gel | Part 2: LEO 43204 Gel 0.075% | Part 2: LEO 43204 Gel 0.1% | Total
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 9 | 32 | 60 | 63 | 224
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 9 | 2 | 3 | 4 | 5 | 3 | 11 | 22 | 23 | 82
  >=65 years | 3 | 10 | 9 | 8 | 7 | 6 | 21 | 38 | 40 | 142
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 6 | 6 | 6 | 6 | 15 | 24 | 26 | 96
  Male | 8 | 9 | 6 | 6 | 6 | 3 | 17 | 36 | 37 | 128
Region of Enrollment [Number; unit: participants]
  Canada | 0 | 0 | 0 | 0 | 0 | 0 | 11 | 20 | 21 | 52
  United States | 12 | 12 | 12 | 12 | 12 | 9 | 21 | 40 | 42 | 172

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Participants Experiencing Dose Limiting Toxicity (DLT) Based on Local Skin Responses (LSRs)
Description: The number participants experiencing a DLT was used to identify the maximum tolerated dose(MTD) levels of LEO 43204 after once daily treatment for 2 consecutive days.The MTD was defined as the highest dose level at which less than 4 out of 12 participants experienced a DLT.
  A DLT was defined as one or more of the following three LSRs:
  * Crusting Grade 4
  * Erosion/Ulceration Grade 4
  * Vesiculation/Pustulation Grade 4
  or two or more of the following five LSRs:
  * Crusting Grade 3
  * Swelling Grade 4
  * Erosion/Ulceration Grade 3
  * Vesiculation/Pustulation Grade 3
  or other clinically relevant signs or symptoms observed, which the Investigator judged to be counted as a DLT.
  The LSRs consists of the following 6 categories: Erythema, flaking/scaling, crusting, swelling, vesiculation/pustulation, erosion/ulceration. Each individual LSR category was given a numeric grade of severity from 0-4. Grade 0 being no presence and Grade 4 being the highest grade of severity.
Time Frame: From Day 1 up to and including Day 8
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: LEO 43204 Gel 0.018% | Part 1: LEO 43204 Gel 0.025% | Part 1: LEO 43204 Gel 0.037% | Part 1: LEO 43204 Gel 0.05% | Part 1: LEO 43204 Gel 0.075% | Part 1: LEO 43204 Gel 0.1%
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 9
Participants
  Yes | 0 | 0 | 2 | 1 | 1 | 0
  No | 12 | 12 | 10 | 11 | 11 | 9

2. Primary Outcome: Part 2: Percent Reduction From Baseline in Actinic Keratosis (AK) Count
Description: Percent reduction from baseline in clinically visible actinic keratosis lesions (AKs) identified in the treatment area.
Time Frame: From baseline to Week 8
Measure: Mean (95% Confidence Interval); unit: percentage of reduction
Arm/Group | Part 2: LEO 43204 Vehicle Gel | Part 2: LEO 43204 Gel 0.075% | Part 2: LEO 43204 Gel 0.1%
Number analyzed (Participants) | 32 | 60 | 63
percentage of reduction | 32.7 [17.9 to 44.8] | 70.0 [64.1 to 74.9] | 62.2 [55.5 to 67.8]
Statistical Analysis 1: Comparison: Part 2: LEO 43204 Vehicle Gel vs Part 2: LEO 43204 Gel 0.075%; Negative binominal regression with log baseline count as offset variable and treatment group and analysis site as factors; Test type: Superiority; p < 0.001, Negative binominal regression; Rate ratio = 0.45, 95% CI 2-sided [0.34 to 0.58]
Statistical Analysis 2: Comparison: Part 2: LEO 43204 Vehicle Gel vs Part 2: LEO 43204 Gel 0.1%; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p < 0.001, Negative binominal regression; Rate ratio = 0.56, 95% CI 2-sided [0.44 to 0.73]
Statistical Analysis 3: Comparison: Part 2: LEO 43204 Gel 0.075% vs Part 2: LEO 43204 Gel 0.1%; Test type: Superiority; p = 0.058, Negative binominal regression; Rate ratio = 1.26, 95% CI 2-sided [0.99 to 1.60]

3. Secondary Outcome: Part 2: Participants With Complete Clearance of AKs (Last Observation Carried Forward [LOCF])
Description: Complete clearance was defined as a 100% reduction from baseline in AK count.
Time Frame: From baseline to Week 8
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: LEO 43204 Vehicle Gel | Part 2: LEO 43204 Gel 0.075% | Part 2: LEO 43204 Gel 0.1%
Number analyzed (Participants) | 32 | 60 | 63
Participants | 3 | 6 | 6
Statistical Analysis 1: Comparison: Part 2: LEO 43204 Vehicle Gel vs Part 2: LEO 43204 Gel 0.075%; Log binomial regression with factors treatment group and baseline AK count as a covariate; Test type: Superiority; p = 0.94, Log binomial regression; Ratio of clearance rates = 1.05, 95% CI 2-sided [0.30 to 4.73]
Statistical Analysis 2: Comparison: Part 2: LEO 43204 Vehicle Gel vs Part 2: LEO 43204 Gel 0.1%; Log binomial regression with factors treatment group and baseline AK count as a covariate; Test type: Superiority; p = 1.00, Log binomial regression; Ratio of clearance rates = 1.00, 95% CI 2-sided [0.28 to 4.51]
Statistical Analysis 3: Comparison: Part 2: LEO 43204 Gel 0.075% vs Part 2: LEO 43204 Gel 0.1%; Log binomial regression with factors treatment group and baseline AK count as a covariate; Test type: Superiority; p = 0.93, Log binomial regression; Ratio of clearance rates = 0.95, 95% CI 2-sided [0.31 to 2.89]

4. Secondary Outcome: Part 2: Participants With Partial Clearance of AKs (LOCF)
Description: Partial clearance was defined as at least 75% reduction from baseline in AK count.
Time Frame: From baseline to Week 8
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: LEO 43204 Vehicle Gel | Part 2: LEO 43204 Gel 0.075% | Part 2: LEO 43204 Gel 0.1%
Number analyzed (Participants) | 32 | 60 | 63
Participants | 5 | 27 | 28
Statistical Analysis 1: Comparison: Part 2: LEO 43204 Vehicle Gel vs Part 2: LEO 43204 Gel 0.075%; Log binomial regression with factors treatment group and baseline AK count as a covariate; Test type: Superiority; p = 0.003, Log binomial regression; Ratio of clearance rates = 2.88, 95% CI 2-sided [1.36 to 7.85]
Statistical Analysis 2: Comparison: Part 2: LEO 43204 Vehicle Gel vs Part 2: LEO 43204 Gel 0.1%; Log binomial regression with factors treatment group and baseline AK count as a covariate; Test type: Superiority; p = 0.004, Log binomial regression; Ratio of clearance rates = 2.84, 95% CI 2-sided [1.35 to 7.74]
Statistical Analysis 3: Comparison: Part 2: LEO 43204 Gel 0.075% vs Part 2: LEO 43204 Gel 0.1%; Log binomial regression with factors treatment group and baseline AK count as a covariate; Test type: Superiority; p = 0.95, Log binomial regression; Ratio of clearance rates = 0.99, 95% CI 2-sided [0.66 to 1.47]

ADVERSE EVENTS:
Time Frame: Part 1: From Day 1 to Week 2 Part 2: From Day 1 to Week 8
Arm/Group | Part 1: LEO 43204 Gel 0.018% | Part 1: LEO 43204 Gel 0.025% | Part 1: LEO 43204 Gel 0.037% | Part 1: LEO 43204 Gel 0.05% | Part 1: LEO 43204 Gel 0.075% | Part 1: LEO 43204 Gel 0.1% | Part 2: LEO 43204 Vehicle Gel | Part 2: LEO 43204 Gel 0.075% | Part 2: LEO 43204 Gel 0.1%
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/9 | 0/32 | 1/60 | 2/63
Other Adverse Events (participants affected / at risk) | 3/12 | 3/12 | 5/12 | 9/12 | 10/12 | 7/9 | 6/32 | 36/60 | 39/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: LEO 43204 Gel 0.018% (N=12) | Part 1: LEO 43204 Gel 0.025% (N=12) | Part 1: LEO 43204 Gel 0.037% (N=12) | Part 1: LEO 43204 Gel 0.05% (N=12) | Part 1: LEO 43204 Gel 0.075% (N=12) | Part 1: LEO 43204 Gel 0.1% (N=9) | Part 2: LEO 43204 Vehicle Gel (N=32) | Part 2: LEO 43204 Gel 0.075% (N=60) | Part 2: LEO 43204 Gel 0.1% (N=63)
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: LEO 43204 Gel 0.018% (N=12) | Part 1: LEO 43204 Gel 0.025% (N=12) | Part 1: LEO 43204 Gel 0.037% (N=12) | Part 1: LEO 43204 Gel 0.05% (N=12) | Part 1: LEO 43204 Gel 0.075% (N=12) | Part 1: LEO 43204 Gel 0.1% (N=9) | Part 2: LEO 43204 Vehicle Gel (N=32) | Part 2: LEO 43204 Gel 0.075% (N=60) | Part 2: LEO 43204 Gel 0.1% (N=63)
Application site pruritus (General disorders) | 2 | 1 | 4 | 7 | 7 | 6 | 1 | 23 | 26
Application site pain (General disorders) | 2 | 1 | 2 | 6 | 6 | 3 | 0 | 15 | 23
Application site paraesthesia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Application site vesicles (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Foreign body reaction (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Administration site reaction (General disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Application site discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Application site inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 3
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Helicobacter gastritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Viral pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nerve compression (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Restless legs syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tension headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin burning sensation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Conjunctivitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eye irritation (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Electrocardiogram qt prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Platelet count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Prostatomegaly (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
LEO acknowledges the investigators right to publish the entire results of the study, irrespective of outcome. LEO retains the right to have any publication submitted to LEO for review. Investigators must undertake not to submit any part of their individual data for publication without the prior consent of LEO.